CLINICAL TRIAL: NCT01179256
Title: Effect of Supplemental Oral Curcumin in Patients With Atopic Asthma
Acronym: CURCUMIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: RICHARD F. LOCKEY, MD, UNIVERSITY OF SOUTH FLORIDA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: curcumin
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Atopic Asthma
Keywords: ASTHMA
MeSH Terms: conditions — Asthma | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CURCUMIN (Experimental): oral supplementation of curcumin 2000mg
  Interventions: Dietary Supplement: CURCUMIN
- PLACEBO (Placebo Comparator): oral PLACEBO TABLET
  Interventions: Other: no intervention other than stopping study

INTERVENTIONS:
Dietary Supplement: CURCUMIN — oral supplementation of curcumin 2000mg
  Arms: CURCUMIN
Other: no intervention other than stopping study — no intervention other than stopping study
  Arms: PLACEBO

SUMMARY:
Curcumin has antioxidant properties and in animal models has numerous molecular targets, many of which are intracellular, such as transcription factors AP-1 and NF. As such, it inhibits the secretion of both pro-inflammatory (TNF-, IL-6) and anti-inflammatory (IL-10) cytokines, possibly by inhibiting transcription factors such as nuclear factor-B (NF-B) and activator protein-1 (AP-1) (Wong et al).

DETAILED DESCRIPTION:
Research Design This is a randomized, double-blinded, placebo-controlled pilot study to evaluate the effects of oral supplementation of curcumin 2000mg, versus placebo, on patients with a history of stable persistent asthma and allergic sensitization.

Ng et al investigated mini-mental status exam (MMSE) scores in 1010 patients without dementia who reported ingesting varying quantities of curry. The authors found a statistically significant improvement in MMSE among patients who reported consuming curry "occasionally", "often, or "very often" (Ng et al). Curcumin is theorized to aid patients with dementia by improving innate immunity and by acting as an anti-inflammatory, antioxidant agent. In a double-blind, placebo-controlled trial of 34 elderly patients with Alzheimer's disease, patients were randomized to receive 0, 1, or 4 grams PO curcumin. While the study did not show significant slowing in cognitive decline over a 6 month period, the dosages were tolerated up to 4 grams without significant adverse effects (Baum et al).

Wong et al demonstrated an inhibitory effect of curcumin on cytokines produced by human cells stimulated by the addition of Dermatophagoides pteronynssinus (Der p1), the major allergen derived from this dust mite. The authors investigated the cytokine changes that occur in bronchial epithelial cells and eosinophils upon activation by Der p1 (increased IL-10, TNF-, IL-6, GM-CSF, and IL-1). Curcumin inhibited such activation. For example, the addition of curcumin decreased the production of IL-10 in Der p1-activated human epithelial/eosinophil co-culture cell lines. Additionally, the addition of curcumin to Der p1-activated eosinophil cell cultures decreased the release of IL-10, TNF-, and IL-1. of NF-B and AP-1 induced by addition of Der p1 in the control group. The authors theorized this occurred via inhibition of AP-1 (Wong et al).

Several additional studies highlight the effect of curcumin in vitro. Curcumin decreases the expression and release of eotaxin, MCP-1, and MCP-3 from IL-1-stimulated human airway smooth muscle cells (Wuyts et al). Additionally, curcumin added to Der f-stimulated lymphocyte cell cultures from allergic asthmatics inhibits Der f-induced lymphocyte proliferation and production of IL-2, IL-4, IL-5, and GM-CSF (Kobayashi et al). Ram et al sensitized guinea pigs with ovalbumin to establish airway hyperresponsiveness. There was a significant decrease in airway constriction and hyperreactivity when curcumin (20mg/kg) was added during the sensitization phase.

There are no clinical studies which have evaluated the effect of oral curcumin supplementation on asthma severity in allergic asthmatics or any in vivo studies in humans with asthma. Therefore, this is a pilot study to evaluate the effects of oral supplementation with curcumin on patients with persistent atopic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-breastfeeding, non-pregnant females
* Aged 18-60 years
* History of physician-diagnosed asthma for 1 year or longer FEV1 60% pre-bronchodilator
* Currently on low or medium dose inhaled corticosteroids (see Appendix 1)
* Use of short-acting β-agonist ≥ 1 in the past 30 days (except for exercise) A ≥ 2+ skin-prick test prick-puncture test to Dermatophagoides pteronyssinus or Dermatophagoidesfarinae with appropriate positive/negative controls (historical is acceptable within 10 years)

Exclusion Criteria:

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Improvement in post-bronchodilator FEV1

SECONDARY OUTCOMES:
Improvement in Asthma Control Test (ACT) Score Decreased frequency of asthma exacerbation
Decreased blood eosinophil count Decreased serum total IgE Decreased in cumulative dose of daily inhaled corticosteroid Decrease serum-specific IgE to Dp and Df Changes in sputum intracellular cytokine profiles (TNF-α, IL-1β, IL-10, IL-4, and IL-5)

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD LOCKEY, MD, Principal Investigator — University of South Florida
Locations (1):
- Usf Asthma Allergy and Immunology Cru, Tampa, Florida, United States